CLINICAL TRIAL: NCT01336595
Title: Comparison of Total Knee Arthroplasties With Oxidized Zirconium and Cobalt Chromium Femoral Components in the Same Patients: A Prospective, Double Blinded, and Randomized Controlled Study
Brief Title: Comparison of Total Knee Arthroplasties With Oxidized Zirconium and Cobalt Chromium Femoral Components
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor and Director, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TKRzirconium
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; oxidized zirconium; genesis II; femoral component; cobalt chrome
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zirconium Femoral Component (Experimental): Oxidized zirconium femoral component of Genesis II TKR system is used.
  Interventions: Device: Zirconium (Zirconium Genesis II)
- Cobalt Chrome (Active Comparator): Cobalt-Chromium Femoral component of Genesis II system is used.
  Interventions: Device: Cobalt-Chrome (Cobalt Chrome Genesis II)

INTERVENTIONS:
Device: Zirconium (Zirconium Genesis II) — Oxidized Zirconium femoral component of Genesis II TKR system is used.
  Other Names: Zirconium Genesis II
  Arms: Zirconium Femoral Component
Device: Cobalt-Chrome (Cobalt Chrome Genesis II) — Cobalt Chrome Femoral Component of Genesis II TKR system is used
  Other Names: Cobalt Chrome Genesis II
  Arms: Cobalt Chrome

SUMMARY:
The purpose of this study is to determine if there are any clinical or radiographic differences in cemented total knee arthroplasty with an oxidized zirconium and a cobalt-chromium femoral knee component.

DETAILED DESCRIPTION:
Although it has been claimed that total knee arthroplasties with an oxidized zirconium femoral knee component had beneficial wear properties in vitro, there are conflicting clinical results. The purpose of the present study was to compare the clinical, subjective, and radiographic results as well as the weight, size and shape of polyethylene wear particles in the patients with an oxidized zirconium and a cobalt-chromium femoral knee component.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2003-01; Primary Completion 2004-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | Initial(one day before surgery), and at 3 months, 1 year, then annually after surgery
  change in knee score will be compared with initial score, until mean follow up of 20 years.

SECONDARY OUTCOMES:
Improvement in the range of motion | Initial(one day before surgery), and at 3 months, 1 year, then annually after surgery
  change in the range of motion of knee joint will be compared with the initial value, until mean follow up of 20 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Won Park, MD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea

REFERENCES:
- [Background] Ezzet KA, Hermida JC, Colwell CW Jr, D'Lima DD. Oxidized zirconium femoral components reduce polyethylene wear in a knee wear simulator. Clin Orthop Relat Res. 2004 Nov;(428):120-4. doi: 10.1097/01.blo.0000148576.70780.13. PMID 15534531
- [Background] Good V, Ries M, Barrack RL, Widding K, Hunter G, Heuer D. Reduced wear with oxidized zirconium femoral heads. J Bone Joint Surg Am. 2003;85-A Suppl 4:105-10. doi: 10.2106/00004623-200300004-00013. No abstract available. PMID 14652400